CLINICAL TRIAL: NCT03001830
Title: GO-8: Gene Therapy for Haemophilia A Using a Novel Serotype 8 Capsid Pseudotyped Adeno-associated Viral Vector Encoding Factor VIII-V3
Brief Title: Gene Therapy for Haemophilia A.
Acronym: GO-8
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL 13/0076; 2016-000925-38 (EudraCT Number); MR/L013185/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2016-12-09; First posted 2016-12-23 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Treatment with AAV2/8-HLP-FVIII-V3
  Interventions: Biological: AAV2/8-HLP-FVIII-V3

INTERVENTIONS:
Biological: AAV2/8-HLP-FVIII-V3 — Infusion of AAV2/8-HLP-FVIII-V3

SUMMARY:
The GO-8 study focuses on assessing safety and efficacy of gene therapy for patients with severe haemophilia A

DETAILED DESCRIPTION:
Haemophilia A is an x-linked, life threatening bleeding disorder arising from defects in the coagulation factor VIII (FVIII) gene. Current treatment for haemophilia A, the commonest inherited bleeding disorder (prevalence of 1 in 5000 individuals) consists of life-long, 2-3 times/week, intravenous injection of clotting factor concentrates, which is demanding and expensive. In contrast, gene therapy offers the potential of a cure for haemophilia A. In a previous gene therapy study in haemophilia B the investigators showed that a single intravenous administration of a serotype 8 based adeno-associated virus, (AAV8) vector encoding the factor IX (FIX) gene resulted in stable (>6 years) therapeutic expression of FIX without long-lasting toxicity. The investigators plan to use the same AAV8 platform to evaluate a novel FVIII expression cassette, AAV2/8-HLP-FVIII-V3, in patient with haemophilia A. Extensive preclinical studies demonstrate that AAV2/8-HLP-FVIII-V3 leads to long-term, endogenous expression of FVIII in mouse and non-human primate models without toxicity even when twenty-fold higher doses than the proposed starting clinical trial dose were used. Therefore, an open label, Phase I/II dose escalation study entailing a single systemic administration of AAV2/8-HLP-FVIII-V3 in adults (>18 years of age) with severe haemophilia A who have baseline factor FVIII levels of <1% of normal has been designed to establish safety and efficacy of our approach. Dosing will begin at 6x10^11 vector genome (vg)/kg progressing sequentially to 2x10^12vg/kg and ultimately 6x10^12vg/kg in the absence of toxicity. A minimum of 2 patients will be recruited at each dose with a possibility of expanding the dose cohort to a maximum of 6 patients based on safety and efficacy. The study duration for each patient will be 5 years after vector infusion.

ELIGIBILITY:
Inclusion criteria:

I. Adult males, ≥ 18 years of age; confirmed diagnosis of severe haemophilia A (baseline plasma hFVIII levels of <1% of normal; assessed by a one-stage clotting or chromogenic assay) II. A severe bleeding phenotype as defined by at least one of the following: (a) On prophylaxis for a history of bleeding or (b) On demand therapy with a current or past history of 4 or more bleeding episodes/year or (c) evidence of chronic haemophilic arthropathy (pain, joint damage, and loss of range of motion) III. Received treatment with hFVIII concentrates with at least >50 exposure days; IV. Able to give full informed consent and able to comply with all requirements of the trial including 5-year long-term follow-up; V. Willing to practice barrier contraception until at least three consecutive semen samples after vector administration are below the sensitivity of the assay for vector sequences.

Exclusion criteria:

VI. Presence of neutralising anti-hFVIII antibodies (inhibitor, determined by the Bethesda inhibitor assay) at the time of enrolment or a previous history of hFVIII inhibitor on at least two occasions that required clinical management ; VII. Use of investigational therapy for haemophilia within 30 days before enrolment; VIII. Subjects with active hepatitis B or C, and HBsAg or hepatitis C RNA viral load positivity, respectively or currently on antiviral therapy for hepatitis B or C. (Negative viral assays in two samples, collected at least six months apart, will be required to be considered negative. Both natural clearers and those who have cleared hepatitis C on antiviral therapy are eligible).

IX. Serological evidence of HIV; X. Evidence of liver dysfunction (persistently elevated alanine transaminase >1.5 times upper limit of normal); XI. Uncontrolled glaucoma, diabetes mellitus, or hypertension (systolic BP consistently ≥140 mmHg or diastolic BP consistently ≥90 mmHg); XII. Any disease or condition (including cancer) at the physician's discretion that would prevent the patient from fully complying with the requirements of the study.; XIII. Suspicious lung lesions on CT scan that raise the possibility of cancer or premalignant pathology (based on chest CT scan done at screening or within 6 months prior to the screening visit) XIV. Presence of liver abnormality that is suspicious of malignancy on screening liver ultrasound XV. Patients with uncontrolled cardiac failure or unstable angina; XVI. Detectable neutralising anti-AAV8 antibodies XVII. Received an AAV vector, or any other gene transfer agent in the previous 6 months except for vaccines XVIII. History of active tuberculosis, fungal disease or other chronic infection XIX. Subjects who are unwilling to provide the required semen samples XX. Poor performance status (WHO score >1) XXI. Patients at high risk of thromboembolic events (high risk patients would include those with a history of arterial or venous thromboembolism (e.g. deep vein thrombosis, pulmonary embolism, non-haemorrhagic stroke, arterial embolus) and those with acquired thrombophilia including conditions such as atrial fibrillation).

XXII. Patients with a CHA2DS2-VASc score of 2 and above

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Safety - Dose Limiting Toxicity possibly attributable to the gene therapy | Up to 5 years post-infusion
  Toxicity will be assessed according to CTCAE, version 4.03 based on the monitoring schedule which comprises a number of clinical and laboratory evaluations
Safety - Neutralising anti-hFVIII antibody development following gene therapy | Up to 5 years post-infusion
  The presence of neutralising hFVIII antibodies will be assessed by regular laboratory tests during patient follow up post infusion

SECONDARY OUTCOMES:
Plasma hFVIII activity | Regularly up to 5 years post-infusion
  Assessments of plasma hFVIII activity
Bleeding frequency | Annual review for 5 years
  Assessment of bleeding frequency using participant diaries before and after gene transfer
hFVIII concentrate usage | Annual review for 5 years
  Assessment of hFVIII concentrate usage as per participant treatment records before and after gene transfer
Immune response to the AAV8 capsid. | Weeks 3, 6, 9 & 12, month 6 and annually post-infusion to Year 5
  Immune response to the AAV8 capsid will be assessed by measurement of the AAV8 antibody titre (humoral response) in plasma samples collected at various time points after gene transfer. Cellular immune response to AAV capsid will be determined using gamma interferon (IFNγ) ELIspot assay to AAV8 capsid
Viral shedding | Weekly from 7 days post infusion until sample clearance.
  Serum and bodily secretions will be collected to assess clearance of vector genomes

CONTACTS AND LOCATIONS:
Overall Officials: Pratima Chowdary, MD, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (4):
- United States (3):
  - St. Luke'S Regional Medical Center, Ltd, Boise, Idaho
  - University of Kentucky, Lexington, Kentucky
  - St Jude's Children's Research Hospital, Memphis, Tennessee
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No